CLINICAL TRIAL: NCT00131118
Title: Efficacy and Safety of Zoledronic Acid in Children (1 -17 Years) With Severe Osteogenesis Imperfecta
Brief Title: Zoledronic Acid in Children (1 -17 Years) With Severe Osteogenesis Imperfecta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446H2202E1
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2016-11

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta, Brittle bone disease, bisphosphonate, children
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
This is an extension study to examine the long-term safety and efficacy of zoledronic acid in patients who have completed the core CZOL446H2202 study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the core CZOL446H2202 study
* Males or females between 1-17 years of age

Exclusion Criteria:

* Deformity or abnormality which would prevent spine bone density from being done
* Any surgical bone-lengthening procedure
* Any kidney diseases or abnormalities
* Low calcium or vitamin D levels in the blood

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Enrollment: 127
Dates: Start 2004-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Long-term safety of two different zoledronic acid doses over an additional 12 months in patients who have completed one year treatment in CZOL446H2202

SECONDARY OUTCOMES:
Measure percentage change of lumbar spine bone mineral density at month 18 and 24 compared to baseline in the core study.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UCLA Medical Center-Dept of Pediatric Nephrology, Los Angeles, California
  - Alfred Dupont Hospital for Children, Wilmington, Delaware
  - Intermountains Orthopedics, Boise, Idaho
  - Children's Hospital, Omaha, Nebraska
  - For information regarding facilities, please contact the Central Contact, Multiple Locations, New Jersey
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: Novartis patient recruitment website — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=371